CLINICAL TRIAL: NCT00130221
Title: Skin Cleansing With Chlorhexidine to Improve Nosocomial Infection Risks. (SCCIN Project)
Brief Title: Skin Cleansing With Chlorhexidine to Decrease Hospital Acquired Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Sage Products, Inc. (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Clinical Research Director, Cook County Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 05-006
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Nosocomial Infection; Bacteremia; Sepsis; Pneumonia; Urinary Tract Infection; Clostridium Infection
Keywords: Chlorhexidine; Blood stream infections; central venous catheter associated; Nosocomial infection; Bacteremia; sepsis; Pneumonia; Urinary tract infection; Clostridium Difficile; intensive care unit; catheter; nosocomial pneumonia; Infection control
MeSH Terms: conditions — Cross Infection; Bacteremia; Sepsis; Pneumonia; Urinary Tract Infections; Clostridium Infections; Healthcare-Associated Pneumonia | interventions — Soaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chlorhexidine gluconate (CHG) (Experimental): daily skin cleansing with no-rinse, 2% CHG-impregnated cloths (Sage)
  Interventions: Drug: 2% chlorhexidine gluconate impregnated cloth
- Soap & Water (Active Comparator): bathing daily with bar soap (Dial Corp., Scottsdale, AZ) warm water, and cotton washcloths
  Interventions: Other: Daily bathing with Bar soap

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate impregnated cloth
  Arms: chlorhexidine gluconate (CHG)
Other: Daily bathing with Bar soap — bathed daily with bar soap (Dial Corp., Scottsdale, AZ), warm water, and cotton washcloths.
  Other Names: Soap
  Arms: Soap & Water

SUMMARY:
Patients in the intensive care unit are at risk for many infections because the severity of illness and the procedures necessary to care for them. This study is designed to look at a change in bathing procedure as a method to reduce infections. Currently, patients at John H. Stroger Hospital are cleansed with soap and water. However, preliminary data from a previous study at Rush University Medical Center showed that a chlorhexidine (CHG)-impregnated cloth (2% CHG Antiseptic Cloth system, Sage Products, Inc.) decreased skin bacteria and may lessen bacteria in the blood stream. The 2% CHG Antiseptic Cloth system is a non-irritating, no-rinse, cleansing and moisturizing product that contains 2% chlorhexidine gluconate. The goal of this proposed study is to further evaluate the effectiveness of the 2% CHG Antiseptic Cloth system compared with soap and water in cleansing the skin and preventing bacteria from entering the bloodstream.

DETAILED DESCRIPTION:
Patients admitted to the medical intensive care unit at John H Stroger Hospital are randomly assigned to Unit A or B. Unit B was randomly selected as the intervention unit. For 6 months, all patients in Unit B will be bathed with the 2% CHG Antiseptic Cloth system and all patients in Unit A will receive soap and water baths. After this 6 month period, there will be a 2 to 4 week washout period and the interventions will cross over, with Unit A receiving Chlorhexidine baths and unit B receiving soap and water for 6 months.

Each week, two randomly selected patients will have cultures of the inguinal area, neck/subclavian region, and endotracheal aspirates. A comparison of the colonization of the skin and sputum will be done between the two intervention groups.

Daily infection surveillance will be done on all patients in the intensive care unit. A comparison of blood stream infections, clinical sepsis, and other nosocomial infections will be done between the two intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Data collection will be compiled from all the participants admitted to the Medical Intensive Care Unit (MICU).
* For skin cultures: One randomly selected (intubated or non-intubated) patient in each intervention group

Exclusion Criteria:

* Patients with greater than 20% of body surface area disruption in skin integrity will be excluded from participation in the 2% CHG Antiseptic Cloths arm of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-07-26 (Actual)

PRIMARY OUTCOMES:
Clinical: Primary blood stream infections and culture negative sepsis | Six Months
  Weekly culture of central line insertion sites
Microbiologic: Skin colonization from environment and endotracheal secretions | Six Months
  Weekly skin cultures

SECONDARY OUTCOMES:
Clinical: Laboratory confirmed blood stream infections | Six months
  Culture positive blood stream infection from patients on investigational units
Nosocomial infections | Six months
  Positive microbiology lab results of Clostridium difficile-associated diarrhea (CDAD), secondary bloodstream infection (BSI), ventilator-associated pneumonia (VAP), urinary tract infection (UTI), and clinical cultures that grew selected resistant bacteria (MRSA, VRE, and A. baumannii).

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Weinstein, MD, Principal Investigator — John H. Stroger Hospital of Cook County
Locations (1):
- John H. Stroger Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Background] Appelgren P, Hellstrom I, Weitzberg E, Soderlund V, Bindslev L, Ransjo U. Risk factors for nosocomial intensive care infection: a long-term prospective analysis. Acta Anaesthesiol Scand. 2001 Jul;45(6):710-9. doi: 10.1034/j.1399-6576.2001.045006710.x. PMID 11421829
- [Background] Beezhold DW, Slaughter S, Hayden MK, Matushek M, Nathan C, Trenholme GM, Weinstein RA. Skin colonization with vancomycin-resistant enterococci among hospitalized patients with bacteremia. Clin Infect Dis. 1997 Apr;24(4):704-6. doi: 10.1093/clind/24.4.704. PMID 9145745
- [Background] Cohen J, Cristofaro P, Carlet J, Opal S. New method of classifying infections in critically ill patients. Crit Care Med. 2004 Jul;32(7):1510-26. doi: 10.1097/01.ccm.0000129973.13104.2d. PMID 15241096
- [Background] Mermel LA, Farr BM, Sherertz RJ, Raad II, O'Grady N, Harris JS, Craven DE; Infectious Diseases Society of America; American College of Critical Care Medicine; Society for Healthcare Epidemiology of America. Guidelines for the management of intravascular catheter-related infections. Clin Infect Dis. 2001 May 1;32(9):1249-72. doi: 10.1086/320001. Epub 2001 Apr 3. No abstract available. PMID 11303260
- [Background] O'grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2002 Dec;30(8):476-89. doi: 10.1067/mic.2002.129427. PMID 12461511
- [Background] Shorr AF, Humphreys CW, Helman DL. New choices for central venous catheters: potential financial implications. Chest. 2003 Jul;124(1):275-84. PMID 12853534
- [Derived] Bleasdale SC, Trick WE, Gonzalez IM, Lyles RD, Hayden MK, Weinstein RA. Effectiveness of chlorhexidine bathing to reduce catheter-associated bloodstream infections in medical intensive care unit patients. Arch Intern Med. 2007 Oct 22;167(19):2073-9. doi: 10.1001/archinte.167.19.2073. PMID 17954801